CLINICAL TRIAL: NCT02842827
Title: A Multi-Center, Open Label Study to Assess the Safety, Steady-State Pharmacokinetics and Pharmacodynamics of IMG-7289 With and Without ATRA (Tretinoin) in Patients With Advanced Myeloid Malignancies
Brief Title: A Study of Bomedemstat (IMG-7289/MK-3543) With and Without ATRA, in Participants With Advanced Myeloid Malignancies (IMG-7289-CTP-101/MK-3543-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMG-7289-CTP-101; IMG-7289-CTP-101 (Other: Imagobio); MK-3543-001 (Other: Merck)
Record Dates: First submitted 2016-07-12; First posted 2016-07-25 (Estimated); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: LSD1; High-risk Acute Myeloid Leukemia; High-risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — bomedemstat; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Cohort 1a: bomedemstat 0.75 mg/kg/day (Experimental): Participants receive bomedemstat 0.75 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat
- Cohort 1b: bomedemstat 1.5 mg/kg/day (Experimental): Participants receive bomedemstat 1.5 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat
- Cohort 1c: bomedemstat 3 mg/kg/day (Experimental): Participants receive bomedemstat 3 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat
- Cohort 1d: bomedemstat 6 mg/kg/day orally (Experimental): Participants receive bomedemstat 6 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat
- Cohort 1x3: bomedemstat 3 mg/kg/day orally plus tretinoin 45 mg/m^2 /day3 (Experimental): Participants receive bomedemstat 3 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat; Drug: tretinoin
- Cohort 1x6: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day (Experimental): Participants receive bomedemstat 6 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants will receive up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
  Interventions: Drug: bomedemstat; Drug: tretinoin
- Cohort 3x: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day (Experimental): Participants receive bomedemstat 6 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 21-day cycles consisting of 14 days of treatment and 7 days of rest. Participants will receive up to 2 cycles (21-day cycles) for up to a total of up 42 days (28 days on treatment).
  Interventions: Drug: bomedemstat; Drug: tretinoin
- Cohort 4x: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day (Experimental): Participants receive bomedemstat 6 mg/kg/day orally for 21 days plus tretinoin 45 mg/m^2/day orally in 28-day cycles consisting of 21 days of treatment and 7 days of rest. Participants will receive at least 1 cycle (28-day cycles) and will receive subsequent cycles at the discretion of the investigator.
  Interventions: Drug: bomedemstat; Drug: tretinoin

INTERVENTIONS:
Drug: bomedemstat — oral administration
  Other Names: MK-3543; IMG-7289
Drug: tretinoin — oral administration
  Other Names: ATRA®; Vesanoid®; all-trans retinoic acid,
  Arms: Cohort 1x3: bomedemstat 3 mg/kg/day orally plus tretinoin 45 mg/m^2 /day3; Cohort 1x6: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day; Cohort 3x: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day; Cohort 4x: bomedemstat 6 mg/kg/day plus tretinoin 45 mg/m^2/day

SUMMARY:
This is an open label study of the dose and duration of an orally administered lysine-specific demethylase 1 (LSD1) inhibitor, bomedemstat, in patients with high-risk acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS). Some participants may also receive all-trans retinoic acid (ATRA; also known as tretinoin and Vesanoid®) in combination with bomedemstat. This study investigates the following:

* The safety and tolerability of bomedemstat with and without ATRA
* The pharmacodynamic effect of different doses of bomedemstat and treatment durations, as well as bomedemstat administered in combination with ATRA
* The pharmacokinetics of bomedemstat with and without ATRA

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

High-risk Acute Myeloid Leukemia (AML)

* Have a diagnosis of AML according to the World Health Organization (WHO) criteria
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score ≤2
* Have AML that is classified as high risk as defined by one of the following: ≥ 60 years of age who were not candidates for or have refused standard chemotherapy; ≥18 years of age with de novo or secondary AML who were not expected to benefit from standard remission-induction chemotherapy; or had relapsed/refractory AML after no more than 3 previous lines of chemotherapy.

High-risk Myelodysplastic Syndromes (MDS)

* Have a diagnosis of myelodysplastic syndromes according to the World Health Organization (WHO) criteria
* Have either an International Prognostic Scoring System (IPSS) score equivalent to intermediate-2 risk or higher, or a Revised International Prognostic Scoring System (IPSS-R) score equivalent to intermediate risk or higher.
* Have MDS that is classified as high risk as defined by one of the following: participants who have failed first-line therapy; or treatment-related MDS, except if it is associated with favorable cytogenetics, and not a candidate for stem cell transplantation
* Prior autologous stem cell transplant is allowed if a minimum of 3 months has elapsed from the time of transplant and the patient has recovered from transplant-associated toxicities
* Prior allogeneic stem cell transplant is allowed, provided all of the following criteria are met: transplant was >120 days prior to study enrollment; no immunosuppressive medications have been taken for at least 1 month; and no active graft versus host disease (GVHD), excluding Grade 1 skin GVHD
* Has a life expectancy >12 weeks

Exclusion Criteria:

* Is receiving other treatments for the condition (with exceptions and time limits)
* Has had major surgery in last 4 weeks or minor surgery in the last 2 weeks
* Has a scheduled hematopoietic stem-cell transplant
* Is currently using prohibited medications
* Has clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia
* Has a concurrent second active and non-stable malignancy
* Has an uncontrolled active infection
* Has known Human Immunodeficiency Virus (HIV) infection or active Hepatitis B or Hepatitis C virus infection
* Has used an investigational agent within last 14 days
* Is a pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1a: Bomedemstat 0.75 mg/kg/Day: Participants received bomedemstat 0.75 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 1b: Bomedemstat 1.5 mg/kg/Day: Participants received bomedemstat 1.5 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 1c: Bomedemstat 3 mg/kg/Day: Participants received bomedemstat 3 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 1d: Bomedemstat 6 mg/kg/Day: Participants received bomedemstat 6 mg/kg/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day: Participants received bomedemstat 3 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day: Participants received bomedemstat 6 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 14-day cycles consisting of 7 days of treatment and 7 days of rest. Participants received up to 4 cycles (14-day cycles) for up to a total of up 56 days (28 days on treatment).
- Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day: Participants received bomedemstat 6 mg/kg/day orally plus tretinoin 45 mg/m^2/day orally in 21-day cycles consisting of 14 days of treatment and 7 days of rest. Participants received up to 2 cycles (21-day cycles) for up to a total of up 42 days (28 days on treatment).
- Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day: Participants received bomedemstat 6 mg/kg/day orally for 21 days plus tretinoin 45 mg/m^2/day orally in 28-day cycles consisting of 21 days of treatment and 7 days of rest. Participants received at least 1 cycle (28-day cycles) and received subsequent cycles at the discretion of the investigator.
Period: Overall Study
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Started | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Treated | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not Completed | 3 | 6 | 4 | 6 | 5 | 8 | 4 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 2 | 3 | 2 | 1 | 0 | 4
Not completed — Physician Decision | 1 | 3 | 0 | 0 | 1 | 4 | 2 | 1
Not completed — Protocol Defined Disease Progression | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant Withdrawal of Consent | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received ≥1 dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Total
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (10.02) | 74.2 (9.24) | 74.0 (10.95) | 66.8 (11.14) | 67.2 (14.65) | 71.8 (9.00) | 68.5 (2.08) | 70.5 (11.65) | 70.6 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4 | 6 | 2 | 3 | 19
  Male | 2 | 5 | 3 | 5 | 1 | 3 | 2 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 4 | 4 | 6 | 4 | 8 | 3 | 6 | 37
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 5 | 4 | 5 | 5 | 7 | 4 | 7 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 5
Disease Diagnosis [Count of Participants; unit: Participants] — A diagnosis of either acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) was a requirement for inclusion in this study.
  Participants
    AML | 2 | 6 | 4 | 6 | 3 | 7 | 4 | 7 | 39
    MDS | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any undesirable physical, psychological, or behavioral effect experienced by a participant during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not related to the study drug. This included any untoward signs or symptoms experienced by the participant from the time of first dose until completion of the study. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 24 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8

2. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE was defined as any adverse event, whether or not related to the study drug, that resulted in any of the following outcomes:
  * Death
  * Life-threatening experience
  * Required or prolonged inpatient hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly
  * Important medical events that, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above.
  The number of participants who experienced an SAE is presented.
Time Frame: Up to approximately 24 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 3 | 6 | 4 | 5 | 5 | 9 | 4 | 8

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any undesirable physical, psychological, or behavioral effect experienced by a participant during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not related to the study drug. This included any untoward signs or symptoms experienced by the participant from the time of first dose until completion of the study. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 18 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 2 | 2 | 3 | 3 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. A DLT was defined as any of the following events that occurs during the DLT evaluation period and is considered by the Investigator possibly, probably, or definitely related to bomedemstat:
  * A clinically significant bleeding event
  * Any Grade 4 or 5 non-haematologic adverse event
  * Any Grade 3 non-haematologic adverse event with failure to recover to Grade 1 within 7 days of drug cessation, with the following exceptions: ≥ Grade 3 nausea, vomiting or diarrhoea that responds to standard medical care and ≥ Grade 3 aesthenia lasting less than 14 days
  * Any Grade 3 electrolyte abnormality unrelated to the underlying malignancy and persisting greater than 24 hours.
  Per protocol, DLTs were measured during the first 28-day treatment period. The number of participants who experienced a DLT is presented.
Time Frame: Up to approximately 28 Days
Population: The DLT population included all participants who received ≥ 1 dose of study treatment and had follow-up through the DLT evaluation period (28 days on treatment) or who discontinued from study treatment due a to drug-related AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Experiencing Any Grade 3 to 5 Adverse Events (AE) as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Description: AEs were graded for severity on a scale of 1 to 5 using CTCAE criteria. Grade 1=mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2=moderate, minimal, local, or noninvasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3=severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care. Grade 4=life-threatening consequences with urgent intervention indicated. Grade 5 =death related to AE. The number of participants who experienced any Grade 3 to 5 AE is reported.
Time Frame: Up to approximately 24 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 3 | 6 | 4 | 5 | 5 | 9 | 4 | 8

6. Primary Outcome: Number of Participants Who Experienced a Medical Event of Interest (MEOI)
Description: Medical Events of Interest (MEOI) were adverse events that did not meet any criteria for a serious adverse event but were of particular interest in the context of the study. MEOIs included bleeding due to low platelets; electrocardiogram (ECG) QT corrected interval prolonged 481-500 milliseconds; and infection where, at a minimum, oral antibiotic, antifungal, or antiviral intervention is indicated. The number of participants with MEOIs is presented.
Time Frame: Up to approximately 24 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9 | 4 | 8
Participants | 1 | 1 | 1 | 2 | 0 | 3 | 0 | 0

7. Primary Outcome: Maximum Concentration (Cmax) of Bomedemstat Alone or Administered With Tretinoin
Description: Cmax was defined as the maximum concentration of bomedemstat observed after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the CMax of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). Unbound plasma concentrations of bomedemstat were estimated by assuming that protein binding was 60.57%. For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the Cmax was determined for participants in Cohort 1. The LOQ of the assay was 1 ng/mL. The Cmax of bomedemstat in unbound plasma is presented.
Time Frame: Cycle 1 Day 1: predose and 1, 2, 3, and 24 hours postdose; Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of Cmax.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9
nanograms/milliliter
  Cycle 1 Day 1 | 10.7 (12.6) | 19.6 (19.0) | 65.7 (22.9) | 145 (85.5) | 66.8 (27.3) | 205 (112)
  Cycle 1 Day 7: number analyzed (Participants) | 2 | 6 | 4 | 6 | 4 | 8
  Cycle 1 Day 7 | 9.67 (12.0) | 18.1 (10.4) | 72.2 (26.0) | 202 (111) | 119 (72.1) | 291 (211)

8. Primary Outcome: Time to Maximum Concentration (Tmax) of Bomedemstat Alone or Administered With Tretinoin
Description: Tmax was the time required to reach the maximum concentration of bomedemstat observed after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the TMax of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the Tmax was determined for participants in Cohort 1. The Tmax of bomedemstat in plasma is presented.
Time Frame: Cycle 1 Day 1: predose and 1, 2, 3, and 24 hours postdose; Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of Tmax.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9
hours
  Cycle 1 Day 1 | 1.00 [0.93 to 3.00] | 2.00 [0.93 to 3.05] | 1.00 [0.92 to 2.08] | 2.06 [1.00 to 3.03] | 1.00 [0.92 to 1.17] | 1.02 [0.97 to 2.50]
  Cycle 1 Day 7: number analyzed (Participants) | 2 | 6 | 4 | 6 | 4 | 8
  Cycle 1 Day 7 | 0.77 [0.53 to 1.00] | 1.50 [0.45 to 3.08] | 1.73 [0.47 to 3.05] | 1.53 [0.53 to 3.08] | 0.50 [0.50 to 0.83] | 0.88 [0.00 to 3.93]

9. Primary Outcome: Area Under the Concentration Time Curve From Time 0 to 24 Hours (AUC0-24hr) Postdose of Bomedemstat Alone or Administered With Tretinoin
Description: AUC0-24hr was defined as the total exposure of bomedemstat over 24 hours after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the AUC 0-24hr of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). Unbound plasma concentrations of bomedemstat were estimated by assuming that protein binding was 60.57%. For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the AUC 0-24hr was determined for participants in Cohort 1. The AUC 0-24hr of bomedemstat in unbound plasma is presented.
Time Frame: Cycle 1 Day 1: predose and 1, 2, 3, and 24 hours postdose; Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of AUC0-24hr.
Measure: Mean (Standard Deviation); unit: hours●nanograms/milliliter
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 9
hours●nanograms/milliliter
  Cycle 1 Day 1 | 26.4 (39.2) | 78.6 (36.8) | 323 (142) | 1361 (789) | 287 (113) | 1138 (621)
  Cycle 1 Day 7: number analyzed (Participants) | 2 | 6 | 4 | 6 | 4 | 8
  Cycle 1 Day 7 | 68.8 (90.4) | 129 (78.0) | 550 (247) | 1361 (747) | 383 (116) | 1702 (1326)

10. Primary Outcome: Elimination Half Life (t1/2) of Bomedemstat Alone or Administered With Tretinoin
Description: t1/2 was the time required to divide the bomedemstat concentration by two after reaching pseudo-equilibrium after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the t1/2 of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the t1/2 was determined for participants in Cohort 1. The t1/2 of bomedemstat in plasma is presented.
Time Frame: Cycle 1 Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of t1/2.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 4 | 2 | 5 | 0 | 3
hours | 130 (NA) — Standard deviation could not be calculated for 1 participant | 103 (23.3) | 103 (8.21) | 110 (49.6) |  | 59.8 (29.4)

11. Primary Outcome: Apparent Total Body Clearance (CL/F) of Bomedemstat Alone or Administered With Tretinoin
Description: CL/F was the volume of plasma from which bomedemstat was eliminated per unit of time after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the CL/F of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the CL/F was determined for participants in Cohort 1. The CL/F of bomedemstat in plasma is presented.
Time Frame: Cycle 1 Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of CL/F.
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 2 | 6 | 4 | 6 | 4 | 7
liters/hour | 5.754 (7.711) | 1.351 (1.246) | 492 (322) | 401 (211) | 472 (88.3) | 287 (131)

12. Primary Outcome: Volume of Distribution (Vz/F) of Bomedemstat Alone or Administered With Tretinoin
Description: Vz/F was the volume of distribution of bomedemstat during the terminal phase after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the Vz/F of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the Vz/F was determined for participants in Cohort 1. The Vz/F of bomedemstat in plasma is presented.
Time Frame: Cycle 1 Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of Vz/F.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 4 | 2 | 5 | 0 | 3
liters | 56354 (NA) — Standard deviation could not be calculated for 1 participant | 224527 (122456) | 99822 (74167) | 63895 (24473) |  | 22539 (6061)

13. Primary Outcome: Terminal Elimination Rate Constant (Kel) of Bomedemstat Alone or Administered With Tretinoin
Description: kel was the rate at which bomedemstat was removed from the body by excretion or metabolism after administration of bomedemstat alone or administered with tretinoin. Plasma samples were collected at multiple time points to estimate the kel of bomedemstat using non-compartmental methods of analysis following oral dosing of participants in Cycle 1 (Cycle 1 = 7 days of treatment and 7 days of rest for a total of 14 days). kel was obtained from the slope of the line, fitted by linear least squares regression, through the terminal points of the log (base e) concentration-time profiles. For the pharmacokinetic analysis, plasma concentrations below the assay limit of quantitation (LOQ) that occurred from predose to the first concentration ≥LOQ were treated as 0 and those that occured thereafter were treated as missing. The LOQ of the assay was 1 ng/mL. Per protocol, the kel was determined for participants in Cohort 1. The kel of bomedemstat in plasma is presented.
Time Frame: Cycle 1 Day 7: predose and 0.5, 1, 2, 3, 4, 8, and 24 hours postdose
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone or administered with tretinoin and who had available data for the analysis of kel.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 4 | 2 | 5 | 0 | 3
1/hour | 0.0053 (NA) — Standard deviation could not be calculated for 1 participant | 0.0071 (0.0020) | 0.0068 (0.0005) | 0.0074 (0.0031) |  | 0.0135 (0.0059)

14. Primary Outcome: Event-free Survival (EFS) For High-risk Acute Myeloid Leukemia (AML) Participants
Description: EFS was defined as the time from the first dose of study treatment to the date of a documented EFS event of resistance, relapse, progression, or death due to any cause as assessed by the investigator. Participants without documented events were censored at the date of the last disease assessment. The EFS, calculated using the Kaplan-Meier method, is presented.
Time Frame: Up to approximately 24 months
Population: All participants with high-risk AML as defined by the protocol, who received ≥1 dose of bomedemstat, had disease assessment at baseline, and had data available for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 2 | 6 | 4 | 6 | 3 | 7 | 4 | 7
Months | 0.87 [0.80 to 0.93] | 0.97 [0.93 to NA] — NA=Upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | 0.93 [0.90 to 18.81] | 2.46 [0.97 to NA] — NA=Upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | 0.93 [0.93 to 3.96] | NA [0.50 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | 1.43 [1.40 to 1.46] | 0.93 [0.47 to 5.59]

15. Primary Outcome: Event-free Survival (EFS) For High-risk Myelodysplastic Syndromes (MDS) Participants
Description: as for outcome 14
Time Frame: Up to approximately 24 months
Population: All participants with high-risk MDS as defined by the protocol, who received ≥1 dose of bomedemstat, had disease assessment at baseline, and had data available for the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Months | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. |  |  |  | 0.75 [0.57 to 0.93] | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. |  | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event.

16. Primary Outcome: Overall Survival (OS) For High-risk Acute Myeloid Leukemia (AML) Participants
Description: OS was defined as the time from the first dose of study treatment until death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up. The OS, calculated using the Kaplan-Meier method, is presented.
Time Frame: Up to approximately 24 months
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 2 | 6 | 4 | 6 | 3 | 7 | 4 | 7
Months | NA [0.80 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. | 18.81 [1.17 to 18.81] | 3.86 [1.07 to NA] — NA=Upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | NA [1.86 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | NA [1.36 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. | NA [0.47 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event.

17. Primary Outcome: Overall Survival (OS) For High-risk Myelodysplastic Syndromes (MDS) Participants
Description: as for outcome 16
Time Frame: Up to approximately 24 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Months | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. |  |  |  | NA [0.57 to NA] — NA=Median and upper confidence interval not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event. |  | NA [NA to NA] — NA=Median and lower and upper confidence intervals not reached at time of data cut-off due to insufficient number of participants with an event.

18. Primary Outcome: Objective Response Rate (ORR) For High-risk Acute Myeloid Leukemia (AML) Participants Determined Using the Revised/Modified International Working Group (IWG) Response Criteria (Cheson et al., 2003) and Assessed by the Investigator
Description: ORR was the percentage of participants with a response of complete remission (CR), CR with incomplete recovery (Cri), morphologic leukaemia-free state (MLFS), partial remission (PR), cytogenetic CR (CRc), molecular CR (CRm), or stable disease (SD):
  * CR: <5% bone marrow (BM) blasts or blasts with Auer rods; no extramedullary disease (EMD); absolute neutrophil count ≥1000/μL; platelets ≥100,000/μL; independent of transfusion
  * Cri: CR with residual neutropenia (<1,000/μL) or thrombocytopenia (<100,000/μL); no EMD; does not require transfusion independence (TI)
  * MLFS: <5% blasts in BM with marrow spicules; no EMD; does not require TI
  * PR: ≥ 50% decrease in BM blasts to a range of 5%-25%; Neutrophils ≥ 1,000/μL; Platelets ≥ 100,000/μL; independent of transfusion. ≤ 5% blasts is PR if Auer rods present
  * CRc: CR+reversion to a normal karyotype if initially abnormal
  * CRm: CR+no evidence of residual disease by molecular testing
  * SD: No evidence of CR, PR, progression, new dysplastic changes
Time Frame: Up to approximately 24 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 2 | 6 | 4 | 6 | 3 | 7 | 4 | 7
Percentage of participants | 50.0 [1.3 to 98.7] | 16.7 [0.4 to 64.1] | 25.0 [0.6 to 80.6] | 50.0 [11.8 to 88.2] | 33.3 [0.8 to 90.6] | 28.6 [3.7 to 71.0] | 0.0 [NA to NA] — NA=No participants achieved an objective response so the 95% confidence interval could not be calculated | 28.6 [3.7 to 71.0]

19. Primary Outcome: Best Overall Response (BOR) For High-risk Acute Myeloid Leukemia (AML) Participants Determined Using the Revised/Modified International Working Group (IWG) Response Criteria (Cheson et al., 2003) and Assessed by the Investigator
Description: BOR was the percentage of participants with a best overall response of CR, Cri, MLFS, PR, CRc, CRm, or SD:
  * CR: <5% bone marrow (BM) blasts or blasts with Auer rods; no extramedullary disease (EMD); absolute neutrophil count ≥1000/μL; platelets ≥100,000/μL; independent of transfusion
  * Cri: CR with residual neutropenia (<1,000/μL) or thrombocytopenia (<100,000/μL); no EMD; does not require transfusion independence (TI)
  * MLFS: <5% blasts in BM with marrow spicules; no EMD; does not require TI
  * PR: ≥ 50% decrease in BM blasts to a range of 5%-25%; Neutrophils ≥ 1,000/μL; Platelets ≥ 100,000/μL; independent of transfusion. ≤ 5% blasts is PR if Auer rods present
  * CRc: CR+reversion to a normal karyotype if initially abnormal
  * CRm: CR+no evidence of residual disease by molecular testing
  * SD: No evidence of CR, PR, progression, new dysplastic changes
Time Frame: Up to approximately 24 months
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 2 | 6 | 4 | 6 | 3 | 7 | 4 | 7
Percentage of participants
  Complete remission (CR) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  CR with incomplete recovery (CRi) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Morphologic leukaemia-free state (MLFS) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Partial remission (PR) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 0.0
  Cytogenetic CR (CRc) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Molecular CR (CRm) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Stable disease (SD) | 50.0 | 16.7 | 25.0 | 50.0 | 33.3 | 14.3 | 0.0 | 28.6

20. Primary Outcome: Objective Response Rate (ORR) For High-risk Myelodysplastic Syndromes (MDS) Participants Determined Using the Revised/Modified International Working Group (IWG) Response Criteria (Cheson et al., 2006) and Assessed by the Investigator
Description: ORR was the percentage of participants with a response of complete remission (CR), partial remission (PR), marrow CR (CRm), cytogenetic response (CyR), or stable disease (SD) lasting for ≥4 weeks:
  * CR: ≤5% myeloblasts in the bone marrow (BM) with normal maturation of all cell lines; persistent dysplasia will be noted; Hgb ≥11 g/dL, Platelets ≥100 X 10^9/L, Neutrophils ≥1.0 X 10^9/L, and 0% Blasts in the peripheral blood
  * PR: All CR criteria if abnormal before treatment except: BM blasts decreased by ≥50% over pretreatment but still >5%. Cellularity and morphology not relevant
  * CRm: ≤ 5% myeloblasts in BM and decrease by ≥50% over pretreatment. Hematological improvement responses in the peripheral blood will be noted in addition to bone marrow CR.
  * CyR: Complete=Disappearance of the chromosomal abnormality without appearance of new ones. Partial= ≥50% reduction of the chromosomal abnormality
  * SD: Failure to achieve at least PR, but no evidence of progression for >8 weeks
Time Frame: Up to approximately 24 months
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Percentage of participants | 100.0 [2.5 to 100.0] |  |  |  | 0.0 [NA to NA] — NA=No participants achieved an objective response so the 95% confidence interval could not be calculated | 0.0 [NA to NA] — NA=No participants achieved an objective response so the 95% confidence interval could not be calculated |  | 0.0 [NA to NA] — NA=No participants achieved an objective response so the 95% confidence interval could not be calculated

21. Primary Outcome: Best Overall Response (BOR) Assessed by the Revised/Modified International Working Group (IWG) Response Criteria (Cheson et al., 2006): High-risk Myelodysplastic Syndromes (MDS) Participants
Description: BOR was the percentage of participants with a best overall response of CR, PR, CRm, CyR, or SD lasting for ≥4 weeks:
  * CR: ≤5% myeloblasts in the bone marrow (BM) with normal maturation of all cell lines; persistent dysplasia will be noted; Hgb ≥11 g/dL, Platelets ≥100 X 10^9/L, Neutrophils ≥1.0 X 10^9/L, and 0% Blasts in the peripheral blood
  * PR: All CR criteria if abnormal before treatment except: BM blasts decreased by ≥50% over pretreatment but still >5%. Cellularity and morphology not relevant
  * CRm: ≤ 5% myeloblasts in BM and decrease by ≥50% over pretreatment. Hematological improvement responses in the peripheral blood will be noted in addition to bone marrow CR.
  * CyR: Complete=Disappearance of the chromosomal abnormality without appearance of new ones. Partial= ≥50% reduction of the chromosomal abnormality
  * SD: Failure to achieve at least PR, but no evidence of progression for >8 weeks
Time Frame: Up to approximately 24 months
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Percentage of participants
  Complete remission (CR) | 0.0 |  |  |  | 0.0 | 0.0 |  | 0.0
  Partial remission (PR) | 0.0 |  |  |  | 0.0 | 0.0 |  | 0.0
  Marrow CR (CRm) | 0.0 |  |  |  | 0.0 | 0.0 |  | 0.0
  Cytogenetic response (CyR) | 0.0 |  |  |  | 0.0 | 0.0 |  | 0.0
  Stable disease (SD) | 100.0 |  |  |  | 0.0 | 0.0 |  | 0.0

22. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in Erythrocyte Count in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in erythrocyte count was measured. Baseline was the erythrocyte count at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in erythrocyte count is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: The analysis population consisted of all participants from Cohort 1 who received ≥1 dose of bomedemstat alone and who had available data for the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6
Percent change | 4.4 (6.66) | 16.7 (19.43) | 17.0 (5.83) | 21.4 (14.97)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.3868, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

23. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in Neutrophil Count in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in neutrophil count was measured. Baseline was the neutrophil count at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in neutrophil count is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 6 | 3 | 6
Percent change | 198.4 (206.33) | 223.3 (259.61) | 198.8 (273.54) | 3218.0 (7780.65)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.7744, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

24. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in Platelet Count in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in platelet count was measured. Baseline was the platelet count at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in platelet count is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6
Percent change | 21.9 (18.15) | 30.4 (73.39) | 313.6 (529.94) | 8.1 (20.79)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.5080, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

25. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in Reticulocyte Count in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in reticulocyte count was measured. Baseline was the reticulocyte count at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in reticulocyte count is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 5 | 4 | 6
Percent change | 47.3 (102.51) | 57.1 (52.48) | 133.5 (158.03) | 26.6 (51.64)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.6109, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

26. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in The Number of Blasts in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in the number of blasts was measured. Baseline was the number of blasts at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in the number of blasts is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 4 | 3 | 6
Percent change | 368.0 (399.54) | 2478.3 (3278.96) | 9.7 (25.23) | 2841.4 (6046.61)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.1151, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

27. Secondary Outcome: Maximum Percent Change From Baseline Up to 28 Days of Treatment in Hemoglobin Level in Whole Blood After Administration of Bomedemstat
Description: Whole blood samples were collected at time intervals during the first 4 cycles (Cycle length = 7 days of treatment and 7 days of rest for a total of 14 days), which corresponds to 28 days on treatment. The percent change from baseline in the hemoglobin level was measured. Baseline was the hemoglobin level at screening or the last available observation prior to the first dose of study drug. An analysis of treatment effect between the doses was determined using a Kruskal-Wallis test. This analysis was done to support the evaluation of plasma concentrations (Cmax and Cmin) and exposure (AUC) on haematopoiesis. Per protocol, the analysis was pre-specified to be done on participants that received bomedemstat alone. The maximum percent change from baseline in hemoglobin level is presented.
Time Frame: Baseline (prior to first dose of study drug) and up to 28 days
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day
Number analyzed (Participants) | 3 | 6 | 4 | 6
Percent change | 1262.1 (429.99) | 476.5 (710.28) | 12.6 (3.76) | 134.4 (296.96)
Statistical Analysis 1: Comparison: Cohort 1a: Bomedemstat 0.75 mg/kg/Day vs Cohort 1b: Bomedemstat 1.5 mg/kg/Day vs Cohort 1c: Bomedemstat 3 mg/kg/Day vs Cohort 1d: Bomedemstat 6 mg/kg/Day; Test type: Other; p = 0.0791, Kruskal-Wallis; p-value of the treatment effect was calculated between all dose arms with ≥3 participants

ADVERSE EVENTS:
Time Frame: Up to approximately 24 months
Description: All-cause mortality was reported on all allocated participants. Serious and non-serious adverse events (AEs) were reported on all participants who received ≥1 dose of study treatment. Progression of underlying malignancy was not reported as an AE if it is consistent with the suspected progression of the underlying cancer.
Arm/Group | Cohort 1a: Bomedemstat 0.75 mg/kg/Day | Cohort 1b: Bomedemstat 1.5 mg/kg/Day | Cohort 1c: Bomedemstat 3 mg/kg/Day | Cohort 1d: Bomedemstat 6 mg/kg/Day | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/6 | 2/4 | 3/6 | 2/5 | 2/9 | 1/4 | 4/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 5/6 | 5/5 | 9/9 | 4/4 | 8/8
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 6/6 | 5/5 | 9/9 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a: Bomedemstat 0.75 mg/kg/Day (N=3) | Cohort 1b: Bomedemstat 1.5 mg/kg/Day (N=6) | Cohort 1c: Bomedemstat 3 mg/kg/Day (N=4) | Cohort 1d: Bomedemstat 6 mg/kg/Day (N=6) | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day (N=5) | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=9) | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=4) | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (7) | 2 (2) | 4 (5) | 1 (1) | 4 (6) | 0 (0) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pantoea agglomerans infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a: Bomedemstat 0.75 mg/kg/Day (N=3) | Cohort 1b: Bomedemstat 1.5 mg/kg/Day (N=6) | Cohort 1c: Bomedemstat 3 mg/kg/Day (N=4) | Cohort 1d: Bomedemstat 6 mg/kg/Day (N=6) | Cohort 1x3: Bomedemstat 3 mg/kg/Day Orally Plus Tretinoin 45 mg/m^2/Day (N=5) | Cohort 1x6: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=9) | Cohort 3x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=4) | Cohort 4x: Bomedemstat 6 mg/kg/Day Plus Tretinoin 45 mg/m^2/Day (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 1 (2) | 2 (3) | 2 (3) | 4 (7) | 1 (1) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 4 (10) | 1 (2) | 3 (5) | 2 (2) | 3 (4) | 1 (1) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Macroglossia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctival oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectropion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (4) | 1 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (7) | 4 (10) | 2 (2) | 1 (4) | 6 (11) | 4 (5) | 7 (10)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (7)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (4) | 2 (4) | 5 (6) | 2 (4) | 7 (9) | 2 (2) | 5 (6)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palatal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (6) | 4 (4) | 2 (4) | 4 (8) | 1 (2) | 5 (6)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site laceration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 4 (6) | 2 (3) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 5 (10)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute haemorrhagic conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Genital injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antiphospholipid antibodies positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma scale abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Inspiratory capacity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary casts (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3) | 3 (5) | 2 (2) | 6 (6) | 2 (2) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 2 (2) | 2 (2)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia differentiation syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 2 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Lead/Coordinating Investigator will have the right to submit for publication any results arising from the study subject to the terms and conditions of the Clinical Trial and Confidentiality Disclosure Agreements.

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT02842827/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT02842827/SAP_001.pdf